CLINICAL TRIAL: NCT03162861
Title: Effects of Lumbar Plexus-sciatic Nerve Block Combined With Sevoflurane on Cognitive Function in Elderly Patients After Hip Arthroplasty: Study Protocol for a Prospective, Single-center, Open-label, Randomized, Controlled, Clinical Trial
Brief Title: Lumbar Plexus-sciatic Nerve Block With Sevoflurane on Cognitive Function in Elderly Patients After Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qinghai University (Other)
Responsible Party: Principal Investigator, Yanhong Guo, Principal Investigator, Qinghai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QinghaiUH_007
Record Dates: First submitted 2017-04-26; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Hip Arthropathy
MeSH Terms: interventions — Anesthesia; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the observation group (Experimental): The elderly patients undergoing unilateral total hip arthroplasty will be randomized to assigned to the observation group. In the observation group, tracheal intubation will be conducted for general anesthesia after lumbar plexus-sciatic nerve block, accompanying sevoflurane inhalation for anesthesia maintenance.
  Interventions: Drug: sevoflurane inhalation for anesthesia
- the control group (Experimental): The elderly patients undergoing unilateral total hip arthroplasty will be randomized to assigned to the control group. In the control group, tracheal intubation will be conducted for general anesthesia, accompanying intravenous administration of propofol for anesthesia maintenance.
  Interventions: Drug: propofol for anesthesia

INTERVENTIONS:
Drug: sevoflurane inhalation for anesthesia — The elderly patients undergoing unilateral total hip arthroplasty will be randomized to assigned to the observation group. In the observation group, tracheal intubation will be conducted for general anesthesia after lumbar plexus-sciatic nerve block, accompanying sevoflurane inhalation for anesthesia maintenance.
  Other Names: sevoflurane group
  Arms: the observation group
Drug: propofol for anesthesia — The elderly patients undergoing unilateral total hip arthroplasty will be randomized to assigned to the control group. In the control group, tracheal intubation will be conducted for general anesthesia, accompanying intravenous administration of propofol for anesthesia maintenance.
  Other Names: propofol group
  Arms: the control group

SUMMARY:
To assume that lumbar plexus-sciatic nerve block combined with sevoflurane can effectively diminish the incidence of cognitive dysfunction in elderly patients after hip arthroplasty.

DETAILED DESCRIPTION:
History and current related studies Elderly patients after total hip arthroplasty often experience postoperative cognitive dysfunction (POCD) and disorders of brain function, such as memories, memory storage and concentration, perception and behavioral disorders. POCD is often transient, can be effectively controlled if measures can be taken timely; otherwise, POCD can become permanent, which may greatly affect the patient's quality of life. At present, pathogenesis and therapeutic effect of POCD are not clear in elderly patients undergoing total hip arthroplasty.

With the help of a nerve stimulator, lumbar plexus combined with sciatic nerve block achieves the precise positioning of the nerve puncture site, and achieves unilateral limb complete anesthesia. The scope of the block is limited, and it has little influence on circulation. Lumbar plexus and sacral sciatic nerve block can effectively suppress stress response to surgery and pain and improve cognitive dysfunction in patients after surgery. Basic fibroblast growth factor (bFGF) has been shown to be associated with cognitive function. The decreased bFGF expression can directly affect the function of nerve cells and cause a decrease in cognitive ability. Sevoflurane can improve cognitive dysfunction after surgery. However, whether sevoflurance can reduce the occurrence of POCD after hip arthroplasty has not been reported.

Adverse events

1. To record adverse events, including incision pain, waist-dorsal muscle pain, spinal cord and nerve injury, hypotension, nausea and vomiting, dyspnea, and bradycardia.
2. If severe adverse events occur, investigators will report details including the date of occurrence and measures taken to treat the adverse events to the principle investigator and the institutional review board within 24 hours.

Data collection, management, analysis, open access

1. Data collection: Case report forms will be collected, processed using Epidata software (Epidata Association, Odense, Denmark), collated, and then recorded electronically by data managers using a double-data entry strategy.
2. Data management: The locked electronic database will be accessible and locked only by the project manager. This arrangement will not be altered. The Affiliated Hospital of Qinghai University, China will preserve all of the data regarding this trial.
3. Data analysis: A professional statistician will statistically analyze the electronic database and will create an outcome analysis report that will be submitted to the lead researchers. An independent data monitoring committee will supervise and manage the trial data, ensuring a scientific and stringent trial that yields accurate and complete data.
4. Data open access: Anonymized trial data will be published at www.figshare.com.

Statistical analysis

1. Statistical analysis will be performed using SPSS 19.0 software (IBM, Armonk, NY, USA) and will follow the intention-to-treat principle.
2. Measurement data will be normally distributed and expressed as the mean ± standard deviation. Count data will be expressed as constituent ratio or rate.
3. bFGF expression, Mini-Mental State Examination (MMSE) score and Montreal Cognitive Assessment (MoCA) score in both groups will be compared using two-sample t-test. Above indexes at three time points in the same group will be will be compared using repeated measures analysis of variance. The incidence of adverse reactions in both groups will be compared using Pearson X2 test.
4. The correlation between serum bFGF expression and cognitive function will be analyzed using Pearson correlation analysis.
5. The significance level will be α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 60-70 years
* American Society of Anesthesiologists (ASA) classification: Class II and class III
* Unilateral hip arthroplasty
* Educational level: Junior high school and above, no cognitive dysfunction before surgery
* Hip joint disease treatment for the first time
* All patients or family members signed the informed consent

Exclusion Criteria:

* Nervous system disease or psychosis
* Allergy to anesthesia
* Poor compliance
* Cardiovascular system disease, severe primary liver and kidney diseases
* Other diseases affecting cognitive function or cognitive dysfunction

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | Change from Baseline Mini-Mental State Examination at 3 day
  To assess cognitive function. Mini-Mental State Examination (MMSE) items include memory, attention and computing ability, orientation, recall ability and language skill. Score range: 0-30. MMSE score < 25 is considered as cognitive dysfunction. All of the above tests will be performed by the same professional attending physician in patients with mental emotional stability.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | day 1 and day 3 after surgery
  To assess cognitive function. Montreal Cognitive Assessment (MoCA) items include execution and visual space function, language expression, attention, naming, delayed recall, abstract thinking, and orientation. Score range: 0-30. MoCA score < 26 is considered as cognitive dysfunction. All of the above tests will be performed by the same professional attending physician in patients with mental emotional stability.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Guo, Ph.D, Principal Investigator — Affiliated Hospital, Qinghai University

IPD SHARING:
Plan to Share IPD: Undecided